CLINICAL TRIAL: NCT01339013
Title: Dead Space Effect of an Anaesthesia Gas Reflector (AnaConDa)
Brief Title: Rebreathing of Carbon Dioxide With a Device Used for Giving Inhalational Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20110322
Record Dates: First submitted 2011-04-13; First posted 2011-04-20 (Estimated); Results first posted 2014-09-11 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Anesthetic Ventilatory Requirements
Keywords: Quantification; ventilatory requirements; charcoal filter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AnaConDa (Active Comparator)
  Interventions: Device: Anesthetic Conserving Device (AnaConDa )

INTERVENTIONS:
Device: Anesthetic Conserving Device (AnaConDa ) — Standard HME was replaced by AnaConDa. AnaConDa has charcoal filter, HME does not.

SUMMARY:
The anesthesia gas reflector (AnaConDa) is built on the adsorptive capacity of active carbon which also adsorbs carbon dioxide in exhaled air. Rebreathing of carbon dioxide thus occurs and must be compensated for by increased ventilation. This study aims at determining how much compensation must be given, based on the hypothesis that rebreathing depends on carbon dioxide level in blood and exhaled air.

ELIGIBILITY:
Inclusion Criteria:

* elective coronary artery by-pass graft surgery
* elective valve replacement surgery
* normal left ventricular ejection fraction on preoperative echocardiography

Exclusion Criteria:

* obstructive lung disease
* restrictive lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Bodelsson, Professor, Principal Investigator — Division of Surgery, Department of Anaesthesia, Skane University Hospital, Lund, Sweden
Locations (1):
- University Hospital, Cardiothoracic Intensive Care, Lund, Sweden

REFERENCES:
- [Result] Sturesson LW, Bodelsson M, Johansson A, Jonson B, Malmkvist G. Apparent dead space with the anesthetic conserving device, AnaConDa(R): a clinical and laboratory investigation. Anesth Analg. 2013 Dec;117(6):1319-24. doi: 10.1213/ANE.0b013e3182a7778e. PMID 24257381

RESULTS

PARTICIPANT FLOW:
Recruitment Details: September 2011 to January 2013, Medical Clinic
Pre-assignment Details: All recruited patients participated uneventfully.
Groups:
- AnaConDa Replaces the Heat and Moisture Exchanger: The conventional Heat and Moisture Exchanger is replaced by the AnaConDa which in turn is replaced by the conventional Heat and Moisture Exchanger.
Period: Overall Study
Arm/Group | AnaConDa Replaces the Heat and Moisture Exchanger
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A total of 6 patients participated. All 6 started with HME, then AnaConDa, finally HME
Groups:
- All Study Participants: Heat and Moisture Exchanger, then AnaConDa, finally Heat and Moisture Exchanger
Arm/Group | All Study Participants
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 63 [58 to 75]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Region of Enrollment [Number; unit: participants]
  Sweden | 6

OUTCOME MEASURES:

1. Primary Outcome: Airway Dead Space With Devices for Heat and Moisture Exchange of Respiratory Gas.
Description: A conventional heat and moisture exchanger used in a respiratory circuit during anasthesia was exchanged by an AnaConDa. The AnaConDa causes re-breathing of carbon dioxide which clinically is equivalent to an increased airway dead space. The total airway dead space effect of the AnaConDa, i.e. volume of the device plus rebreathing from the charcoal filter was measured using the Single Breath Test for carbon dioxide, as was airway deadspace of the conventional Heat and Moisture Exchanger. Airway dead space differences between devices was calculated by subtraction of volumes thus achieved. Difference= Airway dead space AnaConDa - Airway dead space conventional Heat and Moisture Exchanger.
Time Frame: 1 hour
Measure: Median (95% Confidence Interval); unit: mL
Groups:
- AnaConDa: Anesthetic Conserving Device (AnaConDa) has a charcoal filter.
Arm/Group | AnaConDa
Number analyzed (Participants) | 6
mL | 136 [120 to 167]

ADVERSE EVENTS:
Groups:
- AnaConDa: Anesthetic Conserving Device (AnaConDa or ACD) has a charcoal filter.
Arm/Group | AnaConDa
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes